CLINICAL TRIAL: NCT03642210
Title: A Phase 3, Multicenter, Open-Label Study of a Levonorgestrel 52 mg Intrauterine System for the Treatment of Heavy Menstrual Bleeding
Brief Title: Study of a Levonorgestrel 52 mg Intrauterine System for the Treatment of Heavy Menstrual Bleeding
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Medicines360 (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M360-L105
Record Dates: First submitted 2018-08-20; First posted 2018-08-22 (Actual); Results first posted 2024-05-14 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-04

CONDITIONS: Menorrhagia
MeSH Terms: conditions — Menorrhagia | interventions — Levonorgestrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Levonorgestrel 52 mg intrauterine system (Experimental): Levonorgestrel 52 mg intrauterine system, inserted for use up to 6 months
  Interventions: Combination Product: Levonorgestrel 52 mg intrauterine system

INTERVENTIONS:
Combination Product: Levonorgestrel 52 mg intrauterine system — Levonorgestrel 52 mg intrauterine system

SUMMARY:
To assess the efficacy of a levonorgestrel 52 mg intrauterine system as a treatment for heavy menstrual bleeding.

DETAILED DESCRIPTION:
This study is a multicenter, open-label, evaluation of the efficacy and safety of LNG20 IUS for treatment of heavy menstrual bleeding.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Reports subjectively heavy menses for most menses when not using hormonal contraception or a copper IUD
* Healthy females 18-50 years old, inclusive, at the time of enrollment
* Able to read and write, as determined by study personnel
* FSH value ≤30 mIU/mL at screening
* Typical menstrual cycle length of 21-35 days with variation from cycle to cycle of typically 5 days or less
* Has menstrual blood loss in 2 of the 3 cycles during the Screening Phase with ≥ 80 mL per cycle as measured by the AH method
* Uterine sound depth of ≥5.5 cm
* Willing to comply with study visit schedule and assessments, including sanitary product collection and diary completion requirements
* Documented (i.e., printed report) Pap testing, regardless of subject's age, and any indicated evaluation/treatment that demonstrates no need for further evaluation during the course of study participation (i.e., within 10 months after consent)
* Planning to reside within a reasonable driving distance of a research site (approximately 150 miles) for duration of study participation
* Willing to use a medication other than a NSAID as first-line treatment for any pain condition during the duration of study participation
* Willing to abstain from heterosexual intercourse or use acceptable contraception during the screening phase; acceptable contraception includes male or female permanent contraception, withdrawal (if has been using as current method prior to screening) or a barrier method
* If previously pregnant, at least one subjectively heavy menses prior to screening

Exclusion Criteria:

* Currently pregnant
* Planning to attempt to become pregnant during the screening and treatment phases of study participation (i.e., up to approximately 11 months after consent)
* Currently lactating or not having a subjectively heavy menses since discontinuation of lactation prior to screening
* Clinical diagnosis of perimenopause (in the opinion of the investigator) based on one or more of the following: changes in menstrual regularity (e.g., shorter, longer, absent, irregular), hot flashes, sleeping disorder, or changes in mood (e.g., depression, nervous tension, and irritability) within 3 months prior to or during the screening period
* Screening blood laboratory value outside of the normal range that, in the opinion of the investigator, requires treatment or further work-up (i.e., are considered clinically significant)
* Has poor venous access or significant history of inability to have blood samples drawn
* Body habitus or history of lower genital tract abnormalities or prior surgeries which may prohibit proper visualization of the cervix or not allow the uterus to be appropriately instrumented
* History of bicornuate uterus or any other abnormality of the uterus resulting in distortion of the uterine cavity or cervical canal incompatible with insertion
* Prior (documented within 6 months) or baseline study ultrasound examination demonstrating:

  * A congenital or acquired uterine anomaly that distorts the uterine cavity or cervical canal incompatible with insertion;
  * Endometrial polyps (unless previously removed),
  * Fibroids meeting any of the following criteria: Distort the uterine cavity or cervical canal incompatible with insertion; Submucosal location; Exceeding 2 cm in the greatest dimension for any individual fibroid; More than three fibroids of at least 1.5 cm in greatest diameter
  * Clear evidence of adenomyosis consisting of any of the following: Subendometrial cysts; Diffuse adenomyosis based on a heterogeneous myometrial echotexture consisting of Hyperechoic findings (islands of endometrial glands), hypoechoic findings (associated muscle hypertrophy), or "Venetian blind" appearance due to subendometrial echogenic linear striations and acoustic shadowing where endometrial tissues cause a hyperplastic reaction.
* Recently diagnosed or clinically evident cervicitis or upper genital tract infection at the time of IUS insertion (unless successfully treated and considered clinically cured for at least 7 days prior to enrollment)
* History of pelvic actinomycosis infection (i.e., received antibiotic treatment; criterion does not include solely a history of Pap test with actinomyces)
* Postpartum or post-abortion endometritis unless symptoms resolved at least 4 weeks prior to screening
* Chronic endometritis on endometrial biopsy at screening (an endometrial biopsy performed within 6 months of Visit 1 could be used if a report is available with a tissue diagnosis)
* Has any of the following premalignant or malignant diseases:

  * Malignant melanoma
  * Acute malignancies affecting blood or leukemias
  * Gestational trophoblastic disease (unless at least one year with undetectable beta-hCG)
  * Known or suspected cervical, ovarian, vaginal or vulvar cancer
  * Uterine cancer or evidence of uterine malignancy, endometrial intraepithelial neoplasia (EIN) or hyperplasia on an endometrial biopsy at screening (an endometrial biopsy performed within 6 months of Visit 1 could be used if a report is available with a tissue diagnosis)
  * History of breast cancer, or suspicion of breast cancer until proven otherwise
* Has any of the following medical conditions:

  * Bleeding diathesis (inherited or acquired)
  * History of von Willebrand's disease or other known coagulopathy
  * Uncontrolled significant hypertension defined as a sitting systolic blood pressure ≥ 160 mm Hg or diastolic blood pressure ≥ 95 mm Hg at any screening or enrollment visit unless treated and controlled within two weeks of discovery
  * Presence or history of venous thromboembolic diseases (deep vein thrombosis, pulmonary embolism), presence or history of arterial thromboembolic diseases (e.g., myocardial infarction, stroke)
  * Uncontrolled thyroid disorder
  * Sickle cell anemia
  * Diabetes mellitus that is poorly controlled or with end-organ/vascular complications
  * Hyperprolactinemia at screening
  * Acute or severe liver disease or liver tumor
  * Poorly controlled bipolar disorder, schizophrenia, psychosis, major depressive disorder or other major psychiatric disorder according the criteria of the Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-5)
  * History of a positive HIV test or having a partner who is known to be HIV positive
  * Current or history of alcohol, illicit drug or prescription drug abuse within 12 months prior to screening
* Use of antifibrinolytics, platelet aggregation inhibitors, anticoagulants or other similar medications that can increase or decrease bleeding within 30 days prior to and during the screening (EXCEPTION: NSAIDs can be used as second-line treatment for pain management)
* Use of intrauterine or implantable contraception, progestin-only pills, combined hormonal contraceptives or oral progestin therapy within 30 days before screening
* Depomedroxyprogesterone acetate (DMPA) injection within the past 9 months prior to screening (this exclusionary time period can be shortened to 6 months if the subject has also had two spontaneous menstrual cycles [requires minimum of 3 heavy menses] that meet criteria for normal menstrual cycle pattern)
* Use of non-contraceptive estrogen, progesterone, progestin, testosterone, androgen or other gonadotropins (e.g. hCG) within 30 days before screening
* Prior total or partial endometrial ablation or resection
* History of a uterine aspiration or curettage procedure for any indication (other than an office biopsy) within 4 weeks of screening
* Known or suspected allergy to levonorgestrel or hypersensitivity to any component of the product
* Use of an experimental medication or receipt of an experimental treatment for any condition within 30 days of screening
* Study staff or a member of the immediate family of a study staff
* Any condition or circumstance that, in the opinion of the Investigator, would constitute contraindications to participation in the study or would compromise ability to comply with the study protocol, such as any concurrent medical condition that is not stable and well-controlled, that is likely to worsen, or that may require recurrent hospitalizations during study participation

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 105 (Actual)
Dates: Start 2019-01-17 (Actual); Primary Completion 2021-10-12 (Actual); Study Completion 2021-10-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Olariu, MD, PhD, Study Director — COO
Locations (29):
- United States (29):
  - MomDoc Women's Health Research, Scottsdale, Arizona
  - OB/GYN Research, University of California, Davis Health, Sacramento, California
  - Wr-McCr, Llc, San Diego, California
  - Stanford University Medical Center, OB-GYN Clinic, Stanford, California
  - University of Colorado Denver, Aurora, Colorado
  - UF Health Women's Specialists, Jacksonville, Florida
  - Comprehensive Clinical Trials, LLC, West Palm Beach, Florida
  - Emory University School of Medicine, Atlanta, Georgia
  - WR-Mount Vernon Clinical Research, LLC, Sandy Springs, Georgia
  - CR Prime, Idaho Falls, Idaho
  - Johns Hopkins Bayview Medical Center, Baltimore, Maryland
  - University of Michigan Women's Hospital, Ann Arbor, Michigan
  - Washington University in St. Louis School of Medicine, St Louis, Missouri
  - Rex Garn Mabey, Las Vegas, Nevada
  - Women's Health Research Center, Lawrenceville, New Jersey
  - M3 Wake Research, Inc., Raleigh, North Carolina
  - University of Cincinnati Physicians Company, Cincinnati, Ohio
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - The Ohio State University, Columbus, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Magee-Womens Hospital, Center for Family Planning, Pittsburgh, Pennsylvania
  - WR-ClinSearch, LLC, Chattanooga, Tennessee
  - University of Tennessee Medical Center, Knoxville, Tennessee
  - WR-Medical Research Center of Memphis, Memphis, Tennessee
  - Baylor College of Medicine, Houston, Texas
  - University of Utah, Salt Lake City, Utah
  - Eastern Virginia Medical-Conrad Clinical Research Center, Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Creinin MD, Barnhart KT, Gawron LM, Eisenberg D, Mabey RG Jr, Jensen JT. Heavy Menstrual Bleeding Treatment With a Levonorgestrel 52-mg Intrauterine Device. Obstet Gynecol. 2023 May 1;141(5):971-978. doi: 10.1097/AOG.0000000000005137. Epub 2023 Apr 5. PMID 37023455

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 105 eligible women, 18-50 years of age, were enrolled to receive LNG20 IUS. This study did not restrict enrollment based on parity, weight or BMI. Women who did not require contraception (e.g., not heterosexually active, using permanent contraception) were included.
Period: Overall Study
Arm/Group | Levonorgestrel 52 mg Intrauterine System
Started | 105
Modified Intent to Treat (MITT) (MITT: All participants with qualifying Baseline data at study entry for whom the IUS is successfully inserted and for whom there is at least one assessment of MBL during the Treatment Phase Cycle 3 or Cycle 6. All MBL values reported for both validated and unvalidated used feminine hygiene products were included. This is the main population for the efficacy analyses.) | 89
Completed | 81
Not Completed | 24

BASELINE CHARACTERISTICS:
Arm/Group | Levonorgestrel 52 mg Intrauterine System
Number analyzed (Participants) | 105
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.4 (8.3)
Age, Customized [Number; unit: participants]
  Age (years): <35 | 46
  Age (years): ≥35 | 59
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 105
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10
  Not Hispanic or Latino | 95
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 2
  Black or African American | 25
  White | 68
  More than one race | 3
  Unknown or Not Reported | 1
Parity [Count of Participants; unit: Participants]
  Nulliparous | 29
  Parous | 76
BMI (kg/m^2), mean [Mean (Standard Deviation); unit: (kg/m^2)] | 31.1 (9.0)
BMI [Count of Participants; unit: Participants]
  <25 kg/m^2 | 29
  25 - <30 kg/m^2 | 25
  ≥30 kg/m^2 | 51
Current Marital Status [N(%)] [Count of Participants; unit: Participants]
  Never Married | 40
  Married | 48
  Divorced | 12
  Separated | 5
Smoking Status [N(%)] [Count of Participants; unit: Participants]
  Never Smoked | 67
  Ex-Smoker | 18
  Current Smoker | 20
Baseline MBL, Mean [Mean (Standard Deviation); unit: (mL)] | 165.4 (79.1)
Baseline MBL, Median [Median (Full Range); unit: (mL)] | 143.2 [73.4 to 519.7]
BMI (kg/m^2), Median [Median (Full Range); unit: (kg/m^2)] | 29.7 [17.6 to 69.1]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Successful Treatment of Heavy Menstrual Bleeding
Description: Number of participants who completed treatment with an End-of-Treatment menstrual blood loss of <80 ml or ≤50% of baseline
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Levonorgestrel 52 mg Intrauterine System
Number analyzed (Participants) | 89
Participants
  End-of-Treatment MBL < 80 mL | 81
  Decrease in End-of-Treatment MBL to ≤ 50% of Baseline MBL | 83

2. Secondary Outcome: Menstrual Blood Loss - Percent Change From Baseline to Cycle 3 (28 Days Per Cycle; Approximately 3 Months)
Description: • Percent change from Baseline MBL to mid-treatment MBL Cycle 3 (28 days per cycle; approximately 3 months)
Time Frame: 3 months
Measure: Median (Full Range); unit: Percent Change in Absolute MBL (%)
Arm/Group | Levonorgestrel 52 mg Intrauterine System
Number analyzed (Participants) | 85
Percent Change in Absolute MBL (%) | -93.3 [-100.0 to 10.3]

3. Secondary Outcome: Menstrual Blood Loss - Absolute Change in Baseline to Cycle 3 (28 Days Per Cycle; Approximately 3 Months)
Description: • Absolute change in Baseline MBL to mid-treatment MBL Cycle 3 (28 Days Per Cycle; Approximately 3 Months)
Time Frame: 3 months
Measure: Median (Full Range); unit: mL
Arm/Group | Levonorgestrel 52 mg Intrauterine System
Number analyzed (Participants) | 85
mL | -127.8 [-421.4 to 53.8]

4. Secondary Outcome: Menstrual Blood Loss - Absolute Change From Baseline to Cycle 6 (28 Days Per Cycle; Approximately 6 Months)
Description: • Absolute change from Baseline to end-of-treatment MBL Cycle 6 (28 Days Per Cycle; Approximately 6 Months)
Time Frame: 6 months
Measure: Median (Full Range); unit: mL
Arm/Group | Levonorgestrel 52 mg Intrauterine System
Number analyzed (Participants) | 89
mL | -127.0 [-427.6 to 79.7]

5. Secondary Outcome: Menstrual Blood Loss - Percent Change From Baseline to Cycle 6 (28 Days Per Cycle; Approximately 6 Months)
Description: • Percent change from Baseline MBL to end-of-treatment MBL Cycle 6 (28 Days Per Cycle; Approximately 6 Months)
Time Frame: 6 months
Measure: Median (Full Range); unit: Percent Change in Absolute MBL (%)
Arm/Group | Levonorgestrel 52 mg Intrauterine System
Number analyzed (Participants) | 89
Percent Change in Absolute MBL (%) | -97.6 [-100.0 to 57.9]

6. Secondary Outcome: Change in Bleeding/Spotting Days From Baseline, Cycle 3, and Cycle 6.
Description: Number of days bleeding, spotting, and bleeding and/or spotting at Baseline, Cycle 3 (approximately 3 months), and Cycle 6 (approximately 6 months).
Time Frame: 6 months
Measure: Median (Full Range); unit: days
Groups:
- Baseline Bleeding and/or Spotting: Baseline Number of Days with Bleeding and/or Spotting
- Baseline Bleeding Only: Baseline Number of Days with Bleeding Only
- Baseline Spotting Only: Baseline Number of Days with Spotting Only
- Cycle 3 Bleeding and/or Spotting: Cycle 3 Number of Days Bleeding with and/or Spotting
- Cycle 3 Bleeding Only: Cycle 3 Number of Days with Bleeding Only
- Cycle 3 Spotting Only: Cycle 3 Number of Days with Spotting Only
- Cycle 6 Bleeding and/or Spotting: Cycle 6 Number of Days with Bleeding and/or Spotting
- Cycle 6 Bleeding Only: Cycle 6 Number of Days with Bleeding Only
- Cycle 6 Spotting Only: Cycle 6 Number of Days with Spotting Only
Arm/Group | Baseline Bleeding and/or Spotting | Baseline Bleeding Only | Baseline Spotting Only | Cycle 3 Bleeding and/or Spotting | Cycle 3 Bleeding Only | Cycle 3 Spotting Only | Cycle 6 Bleeding and/or Spotting | Cycle 6 Bleeding Only | Cycle 6 Spotting Only
Number analyzed (Participants) | 87 | 87 | 87 | 88 | 88 | 88 | 79 | 79 | 79
days | 6.5 [3.6 to 13.0] | 4.5 [2.0 to 11.0] | 1.5 [0.0 to 5.3] | 9.0 [0.0 to 28.0] | 3.0 [0.0 to 20.0] | 5.5 [0.0 to 28.0] | 6.0 [0.0 to 28.0] | 1.0 [0.0 to 25.0] | 3.0 [0.0 to 25.0]

7. Secondary Outcome: Blood Changes - Hemoglobin
Description: • Percent change in hemoglobin from Baseline to mid-treatment (approximately 3 months), from Baseline to end-of-treatment (approximately 6 months), and from mid-treatment to end-of-treatment (approximately 3 months).
Time Frame: 6 months
Measure: Median (Full Range); unit: % change of hemoglobin (g/dL)
Groups:
- Percentage Change From Baseline to Mid-Treatment (Visit 7): Percentage Change in hemoglobin from Baseline to Mid-Treatment (Visit 7)
- Percentage Change From Baseline to End of Treatment (Visit 8): Percentage Change in hemoglobin from Baseline to End of Treatment (Visit 8)
- Percentage Change From Mid-Treatment (Visit 7) to End of Treatment (Visit 8): Percentage Change in hemoglobin from Mid-Treatment (Visit 7) to End of Treatment (Visit 8)
Arm/Group | Percentage Change From Baseline to Mid-Treatment (Visit 7) | Percentage Change From Baseline to End of Treatment (Visit 8) | Percentage Change From Mid-Treatment (Visit 7) to End of Treatment (Visit 8)
Number analyzed (Participants) | 92 | 79 | 76
% change of hemoglobin (g/dL) | 3.5 [-55.6 to 89.9] | 5.5 [-11.0 to 42.1] | 3.9 [-15.0 to 123.6]

8. Secondary Outcome: Blood Changes - Hematocrit
Description: • Percent change in hematocrit from Baseline to mid-treatment (approximately 3 months), from Baseline to end-of-treatment (approximately 6 months), and from mid-treatment to end-of-treatment (approximately 3 months).
Time Frame: 6 months
Measure: Median (Full Range); unit: Hematocrit %
Groups:
- Percentage Change From Baseline to Mid-Treatment (Visit 7): Percentage Change in hematocrit from Baseline to Mid-Treatment (Visit 7)
- Percentage Change From Baseline to End of Treatment (Visit 8): Percentage Change in hematocrit from Baseline to End of Treatment (Visit 8)
- Percentage Change From Mid-Treatment (Visit 7) to End of Treatment (Visit 8): Percentage Change in hematocrit from Mid-Treatment (Visit 7) to End of Treatment (Visit 8)
Arm/Group | Percentage Change From Baseline to Mid-Treatment (Visit 7) | Percentage Change From Baseline to End of Treatment (Visit 8) | Percentage Change From Mid-Treatment (Visit 7) to End of Treatment (Visit 8)
Number analyzed (Participants) | 92 | 81 | 78
Hematocrit % | 2.5 [-12.8 to 57.5] | 4.5 [-12.4 to 32.2] | 2.2 [-16.9 to 27.3]

9. Secondary Outcome: Blood Changes - Ferritin
Description: Change in serum ferritin from Baseline to mid-treatment (approximately 3 months) and to end-of-treatment (approximately 6 months).
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Baseline Ferritin: baseline ferritin (ng/mL)
- Mid-Treatment Ferritin: mid-treatment ferritin (ng/mL)
- End-of-Treatment Ferritin: end-of-treatment ferritin (ng/mL)
Arm/Group | Baseline Ferritin | Mid-Treatment Ferritin | End-of-Treatment Ferritin
Number analyzed (Participants) | 105 | 92 | 82
ng/mL | 30.2 (154.5) | 19.0 (18.1) | 22.4 (17.6)

10. Secondary Outcome: Number of Participants That Discontinued vs Completed Full Treatment Duration
Description: Number of Participants that Discontinued vs Completed Full Treatment Duration.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Levonorgestrel 52 mg Intrauterine System
Number analyzed (Participants) | 105
Participants
  Safety Population | 105
  Discontinued After Failed Insertion | 0
  Completed Full Treatment Duration | 82
  Early Discontinuation | 23

11. Secondary Outcome: Participant Subjective Assessments
Description: • Subjective assessment of menstrual bleeding changes based on VAS questionnaires of Safety and Continuation Rates from Baseline to Treatment Cycle 3 (approximately 3 months) to Cycle 6 (approximately 6 months). Participants responded to various questions regarding their menstrual bleeding on Visual Analog Scales (VAS), with "Not Acceptable" at 0 cm and "Completely Acceptable" at 10 cm.
Time Frame: 6 months
Measure: Median (Full Range); unit: score on a scale in cm
Groups:
- Baseline (Median): At Baseline (Median)
- Cycle 3 (Mid-Treatment) (Median): At Cycle 3 (Mid-Treatment) (Median)
- Cycle 6 (End-of-Treatment) (Median): At Cycle 6 (End-of-Treatment) (Median)
Arm/Group | Baseline (Median) | Cycle 3 (Mid-Treatment) (Median) | Cycle 6 (End-of-Treatment) (Median)
Number analyzed (Participants) | 89 | 89 | 89
score on a scale in cm
  How heavy was your bleeding? (10 cm = worst) | 8.2 [5.9 to 10.0] | 1.9 [0.0 to 7.0] | 1.0 [0.0 to 6.6]
  How acceptable was your bleeding? (0 cm = worst) | 1.8 [0.0 to 9.8] | 8.7 [0.0 to 10.0] | 9.2 [0.0 to 10.0]
  How much cramping pain did you have? (10 cm = worst) | 6.3 [0.0 to 10.0] | 1.4 [0.0 to 7.7] | 0.8 [0.0 to 10.0]
  How much did it interfere with your ability to do daily activities? (10 cm = worst) | 6.2 [0.6 to 9.7] | 0.5 [0.0 to 8.0] | 0.2 [0.0 to 10.0]
  How much did it affect your ability to sleep? (10 cm = worst) | 5.3 [0.0 to 9.6] | 0.3 [0.0 to 3.9] | 0.2 [0.0 to 10.0]

12. Secondary Outcome: Changes in Number of Bleeding Episodes
Description: • Changes from Baseline to mid-treatment Cycle 3 (approximately 3 months), from Baseline to end of treatment Cycle 6 (approximately 6 months), and from mid-treatment Cycle 3 to end of treatment Cycle 6 in the number of bleeding episodes. Bleeding episodes are defined as all bleeding days separated by no more than one bleeding-free day.
Time Frame: 6 months
Measure: Median (Full Range); unit: Bleeding Episodes
Groups:
- Change From Baseline to Treatment Cycles 3: Change from Baseline to Treatment Cycles 3 in total number of bleeding episodes
- Change From Baseline to Treatment Cycles 6: Change from Baseline to Treatment Cycles 6 in total number of bleeding episodes
- Change From Treatment Cycle 3 to Treatment Cycle 6: Change from Treatment Cycle 3 to Treatment Cycle 6 in total number of bleeding episodes
Arm/Group | Change From Baseline to Treatment Cycles 3 | Change From Baseline to Treatment Cycles 6 | Change From Treatment Cycle 3 to Treatment Cycle 6
Number analyzed (Participants) | 87 | 78 | 79
Bleeding Episodes | 0 [-1.5 to 2.5] | -0.9 [-1.5 to 1.5] | 0 [-3.0 to 1.0]

ADVERSE EVENTS:
Time Frame: 6 months
Description: An Adverse Event (AE) was defined as any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment. An AE could be any unfavorable and unintended sign (including a clinically significant abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.
Arm/Group | Levonorgestrel 52 mg Intrauterine System
All-Cause Mortality (participants affected / at risk) | 0/105
Serious Adverse Events (participants affected / at risk) | 0/105
Other Adverse Events (participants affected / at risk) | 49/105
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Levonorgestrel 52 mg Intrauterine System (N=105)
Nausea (Gastrointestinal disorders) | 3 (3)
Bacterial vaginosis (Infections and infestations) | 9 (9)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 3 (3)
Procedural pain (Injury, poisoning and procedural complications) | 2 (2)
Device expulsion (Product Issues) | 9 (9)
Pelvic pain (Reproductive system and breast disorders) | 4 (4)
Vaginal discharge (Reproductive system and breast disorders) | 3 (3)
Acne (Skin and subcutaneous tissue disorders) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 2 (2)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 2 (2)
Nasopharyngitis (Infections and infestations) | 2 (3)
Pneumonia (Infections and infestations) | 2 (2)
Urinary tract infection (Infections and infestations) | 2 (2)
Vulvovaginal mycotic infection (Infections and infestations) | 2 (2)
Headache (Nervous system disorders) | 2 (2)
Dysmenorrhoea (Reproductive system and breast disorders) | 2 (2)
Metrorrhagia (Reproductive system and breast disorders) | 2 (2)
Uterine spasm (Reproductive system and breast disorders) | 2 (2)
Vaginal odour (Reproductive system and breast disorders) | 2 (2)
Vulvovaginal pruritus (Reproductive system and breast disorders) | 2 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2020-02-05): https://cdn.clinicaltrials.gov/large-docs/10/NCT03642210/Prot_000.pdf
  • Statistical Analysis Plan (2021-10-18): https://cdn.clinicaltrials.gov/large-docs/10/NCT03642210/SAP_001.pdf